CLINICAL TRIAL: NCT01907620
Title: Circulating Oxidative Stress and Gestational Hypertension. Study of the Evolution of Free-radical Markers of Oxidative Stress From Before to After Childbirth in Two Groups of Women: Normal Pregnancy and Pre-eclampsia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple
Other Study IDs: Sagot PHRC IR 2007
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Pregnancy Complicated by Pre-eclampsia.; Normal Pregnancy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Normal pregnancy (Other): women pregnant
  Interventions: Other: blood sample
- pregnancy complicated by pre-eclampsia (Other): women with pregnancy complicated by pre-eclampsia
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
The aim of this study is to explore a mechanism that could potentially explain why women with a pregnancy complicated by pre-eclampsia are described as having an increased risk of cardiovascular disease later in life.

If the hypothesis of this study turns out to be true, that is to say that women with pre-eclampsia have a higher level of oxidative stress than women with a normal pregnancy and that this difference persists after the delivery (6 months), a controlled randomized interventional study aiming to evaluate either therapeutic supplementation with antioxidant vitamins (Vit C and E) or modifications in diet could be envisaged.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided written informed consent
* Patients covered by a Health Insurance scheme
* Age > 18 years
* Normal pregnancy
* or pre-eclampsia defined according to the following classical criteria: (i) de novo hypertension defined by arterial blood pressure of at least 140 mm Hg (systolic) or at least 90 mm Hg (diastolic) confirmed by at least two measurements separated by at least 4-6 h, occurring after the 20th week of gestation in a women known beforehand to have a normal blood pressure, (ii) proteinuria defined by urinary excretion of at least 300 mg of protein per 24 h. If 24-hour urine is not available, proteinuria is defined as a concentration of urinary protein of 300 mg/L or more (or >1 + on the urinary dip) in at least two samples of urine taken randomly, but at an interval of at least 4-6 h [7]. Pre-eclampsia is defined as severe if: persistent systolic BP > 170 mm Hg and/or diastolic BP > 110 mm Hg, and/or diuresis < 30 ml/hour, and/or at least 2 of the following signs (headache, phosphenes, epigastric pain or vomiting, pyramidal-type patellar reflexes, papilledema, hepatic pain, thrombopenia < 100x106 /l, ALT AST > 70 UI/l and or hemolysis manifesting as haptoglobin < 0.06 g/l, or a fall in LDH or the presence of schistocytes, the latter three signs define the HELLP syndrome) and/or seizures.
* Term> 26 SA.

Exclusion Criteria:

* Refusal to provide consent
* Context of patent infection.
* Premature rupture of the fetal membranes.
* preexisting or gestational diabetes.
* Vasculoplacental diseases other than pre-eclampsia: placental abruption or infarction, intrauterine growth retardation of in utero fetal death not occurring in a context of pre-eclampsia.
* Chronic or gestational AHT not meeting the criteria for pre-eclampsia.
* Twin/multiple pregnancies

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
quantification of radical species | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Dijon, Dijon, France